CLINICAL TRIAL: NCT06137248
Title: Randomized Study to Assess Colonic Microbiota Changes in Response to Energy Drink Consumption
Brief Title: Study to Assess Colonic Microbiota Changes in Response to Energy Drink Consumption
Acronym: ROSANNA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: McJunkin Family Charitable Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UF-CCPS-037; OCR43110 (Other: University of Florida); IRB202301911 (Other: University of Florida)
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer
Keywords: energy drink; sulfur; taurine; colorectal cancer; microbiota
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Energy Drinks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Energy drink intervention (Experimental)
  Interventions: Dietary Supplement: Energy drink
- Control arm (No Intervention): Participants on this arm will only consume their normal diet for 4 weeks.

INTERVENTIONS:
Dietary Supplement: Energy drink — Participants on this arm will consume an energy drink once daily in addition to their normal diet for 4 weeks.
  Arms: Energy drink intervention

SUMMARY:
This study will investigate whether short-term daily energy drink consumption results in an increase in hydrogen sulfide-producing bacteria in adults 18-40 years old.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the 2nd leading cause of cancer deaths in the US. The bulk of new diagnoses typically occurs after the age of 50 for those without personal or family histories of this disease. However, rates of colorectal cancer have been slowly increasing in incidence in those younger than 50, recently prompting the U.S. Preventative Services Task Force to recommend reducing the age of routine screening to 45. The reason for the rising incidence of CRC in younger individuals (eoCRC) is unclear but with many speculative causes postulated. One of the most frequently cited possible causes relates to changes in the young adult colonic microbiome which either removes a protective mechanism or promotes a carcinogenic process. The latter is the hypothesis being persued.

Certain commensal bacteria produce hydrogen sulfide (H2S) during fermentation of sulfate containing compounds such as sulfur amino acids. For example, Fusobacterium nucleatum produces H2S from metabolizing methionine and cysteine. Atopobium parvulum is another potent H2S producer and is implicated in halitosis. Importantly, H2S has the capacity to induce inflammation and possesses genotoxic and potentially pro-tumorigenic properties, particularly when consistently present over a prolonged period of time. While Fusobacterium and Atopobium are minor members of the normal gut microbiota, recent studies showed that they are overrepresented in CRC patients. The invvestigators published that the relative abundance of A. parvulum was positively correlated with the severity of pediatric inflammatory bowel disease (IBD). Moreover, the investigators observed that Il10-/- mice colonized by A. parvulum developed severe colitis, which was attenuated by a chow diet containing the H2S scavenger bismuth. Together, this data suggests that bacteria-derived H2S may contribute to intestinal pathologies including the creation of a pro-inflammatory and pro-carcinogenic environment, which could be modulated by availability of dietary sulfur contents.

One major energy source for H2S producing gut microbiota is taurine, an essential amino acid found in very high levels/concentrations in energy drinks. The typical American diet provides between 123 and 178 mg of taurine daily. However, consumption of one 8-oz energy drink can increase the average taurine intake 6 to 16 times that our regular diet. The hypothesis being persued is that energy-drinks, through their high taurine content, favors expansion of already present bacteria producing H2S, thereby representing an association with a carcinogenic risk-factor that might help explain the rise in eoCRC cases and developing future interventions to mitigate this risk.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age AND ≤ 40 years of age
* Written informed consent obtained from the subject and the subject agrees to comply with all the study-related procedures
* Subject willing to complete/comply with study required specimen and survey assessments
* Current energy drink consumption of ≤2 energy drinks weekly
* Written informed consent obtained from the subject to participate in two companion biobanks: 1) Dr. Thomas George's Tumor and Biospecimen Sample Biobank and 2) Dr. Ryan Thomas's Microbiorepository for future research.

Exclusion Criteria:

* Personal history of colorectal cancer (CRC)
* Inflammatory Bowel Disease (IBD)
* Chronic diarrhea or other chronic gastrointestinal (GI) problems felt to interfere with study conduct per the PI
* Regular (daily) intake of probiotics
* Oral or IV antibiotic use within the past 28 days (prior to intervention start date)
* Known intolerance of or sensitivity to caffeine
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.
* Known pregnancy at the time of enrollment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
Change in the hydrogen sulfide-metabolizing species of bacteria | 4 weeks
  Determine the change in the hydrogen sulfide-metabolizing species of bacteria in those receiving the energy drink intervention compared to the control group, as measured by the change from baseline to 1 month post-intervention in the sulfur-metabolizing bacterial communities value in the stool

SECONDARY OUTCOMES:
Changes in colonic microbiota | 4 weeks
  Determine changes to the colonic microbiota in participant stool samples between baseline and study completion and associated subject demographic differences and dietary intake
Microbiome changes | 4 weeks
  Determine the concordance of microbiome changes in participant stool samples with dietary logs
Overall change in microbial diversity | 4 weeks
  Determine overall change in microbial diversity in participant stool between baseline and study completion as measured by change in alpha diversity
Overall change in microbial diversity | 4 weeks
  Determine overall change in microbial diversity in participant stool between baseline and study completion as measured by change in Shannon diversity index
Microbiome changes and tolerance | 4 weeks
  Determine subgroup analyses between the two arms regarding microbiome changes and tolerance with regards to gender, race, ethnicity, and baseline dietary meat/seafood/energy drink consumption

CONTACTS AND LOCATIONS:
Overall Officials: Thomas George, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States